CLINICAL TRIAL: NCT01299350
Title: Randomized Comparison Between Nt-proBNP or Clinical Guided Discharges in Patients Hospitalized With Acute Heart Failure
Brief Title: Nt-proBNP Versus Clinical Guided Discharge in Acute Heart Failure
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Juan Sanchis, Full Professor of Medicina, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: University of Valencia
Record Dates: First submitted 2011-02-17; First posted 2011-02-18 (Estimated); Last update posted 2014-04-10 (Estimated); Status verified 2014-04

CONDITIONS: Heart Failure
Keywords: Heart failure; Nt-proBNP
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual (No Intervention): Every patient will receive the drug treatment indicated in the guidelines of the European Society of Cardiology. Patients will be discharged according to routine clinical practice based on symptoms, physical examination and other data that the cardiologist deems appropriate, except for Nt-proBNP.
- Nt-proBNP guided (Experimental): Every patient will receive the drug treatment indicated in the guidelines of the European Society of Cardiology. Patients will be discharged the third day if NT-proBNP levels drops >30% compared to admission values. If such a reduction is not achieved, then the pharmacological treatment will be increased and NT-proBNP will be measured the following days until reaching the 30% reduction. The cutoff point of 30% reduction in NTproBNP was chosen based on previous studies
  Interventions: Other: Nt-proBNP guided discharge

INTERVENTIONS:
Other: Nt-proBNP guided discharge — Every patient will receive the drug treatment indicated in the guidelines of the European Society of Cardiology. Patients will be discharged the third day if NT-proBNP levels drops >30% compared to admission values. If such a reduction is not achieved, then the pharmacological treatment will be increased and NT-proBNP will be measured the following days until reaching the 30% reduction. The cutoff point of 30% reduction in NTproBNP was chosen based on previous studies
  Arms: Nt-proBNP guided

SUMMARY:
Our objective is to compare a policy of hospital discharge guided by NT-proBNP levels versus discharge guided by conventional clinical criteria, in patients admitted with acute heart failure. The hypothesis is that the Nt-proBNP guided discharge will shorten hospital stay without worsening the outcome

DETAILED DESCRIPTION:
Nt-proBNP levels as well as their response to pharmacological treatment are predictive of prognosis in patients with heart failure. The purpose of the present project is to investigate, in patients hospitalized with acute heart failure, whether a discharge decision guided by Nt-proBNP response shortens hospital stay and improves prognosis The included patients will be randomly assigned to one of these two strategies: hospital discharge according to clinical conventional criteria or discharge guided by Nt-proBNP. All patients will be treated following clinical guidelines. In the guided Nt-proBNP strategy, patients will be discharged the third day if NT-proBNP levels drops >30% compared to admission values. If such a reduction is not achieved, then the pharmacological treatment will be increased and NT-proBNP will be measured the following days until reaching the 30% reduction. In the conventional strategy, patients will be discharged at criterion of the attending cardiologist according to clinical assessment without Nt-proBNP. The main outcome will be the number of days of hospitalization at the index episode, and the secondary outcome will be death or readmission by heart failure at one and 6 months. Our hypothesis is that the Nt-proBNP guided discharge will allow to precisely evaluate the response to treatment and to determine the best time for hospital discharge. This will reduce hospital stay and death or readmission rate after discharge.

ELIGIBILITY:
Inclusion Criteria:

1. clinical signs and symptoms of acute heart failure, according to the criteria of the European guidelines
2. NT-proBNP levels > 1000 pg/ml at the time of admission
3. age over 18 years old
4. signed informed consent

Exclusion Criteria:

1. GFR less than 30 ml/minute/m2,
2. life expectancy as determined by concomitant diseases under one year,
3. acute coronary syndrome within 10 days prior,
4. valvular heart disease with surgical approach,
5. infection or process active malignancy,
6. chronic respiratory failure with pulmonary disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2010-11; Primary Completion 2012-10 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Days of hospitalization | At the index episode (at discharge)

SECONDARY OUTCOMES:
Death or readmission by heart failure | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clínico Universitario, Valencia, Valencia, Spain